CLINICAL TRIAL: NCT03956602
Title: Effects of Snack Types on Acute Glucose and Insulin Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HS-2019-0094
Record Dates: First submitted 2019-04-25; First posted 2019-05-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Satiety
MeSH Terms: interventions — Mangifera indica extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Pretzels (Active Comparator): Subjects consume pretzels to examine postprandial response
  Interventions: Other: Pretzels
- Brazil nuts (Experimental): Subjects consume Brazil nuts to examine postprandial response
  Interventions: Other: Brazil nuts
- Potato chips (Active Comparator): Subjects consume potato chips to examine postprandial response
  Interventions: Other: Potato chips
- Mixed nuts (Experimental): Subjects consume mixed nuts to examine postprandial response
  Interventions: Other: Mixed nuts
- White bread (Active Comparator): Subjects consume white bread to examine postprandial response
  Interventions: Other: White bread
- Dried mango (Experimental): Subjects consume dried mango to examine postprandial response
  Interventions: Other: Dried mango
- Mango fruit (Experimental): Subjects consume fresh mango to examine postprandial response
  Interventions: Other: Mango fruit

INTERVENTIONS:
Other: Pretzels — To examine postprandial responses of pretzel consumption
  Arms: Pretzels
Other: Brazil nuts — To examine postprandial responses of Brazil nut consumption
  Arms: Brazil nuts
Other: Potato chips — To examine postprandial responses of potato chip consumption
  Arms: Potato chips
Other: Mixed nuts — To examine postprandial responses of mixed nut consumption
  Arms: Mixed nuts
Other: White bread — To examine postprandial responses of white bread consumption
  Arms: White bread
Other: Dried mango — To examine postprandial responses of dried mango consumption
  Arms: Dried mango
Other: Mango fruit — To examine postprandial responses of fresh mango consumption
  Arms: Mango fruit

SUMMARY:
The purpose of the present study was to determine the effects of different type of snack consumption on postprandial satiety, glucose, insulin, antioxidant capacity and anxiety in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old

Exclusion Criteria:

* Smoker
* Pregnant woman
* Required dietary supplement use
* Required medication of metabolic disorders
* Allergy to nuts or gluten (wheat)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change of Satiety | 0, 20, 40, 60, 90 and 120 minutes post snack consumption
  Hunger feeling (appetite) will be examined using visual analog scale (0-10): 0 least and 10 greatest
Change of glucose level | 0 and 40 minutes post snack consumption
  Blood will be collected by finger pricks and change of glucose level will be examined.
Change of insulin level | 0 and 40 minutes post snack consumption
  Blood will be collected by finger pricks and change of insulin level will be examined
Change of anxiety feeling | 0 and 40 minutes post snack consumption
  Anxiety feeling will examined using STAI (Spielberger Stasumte-Trait Anxiety Inventory) questionnaire (1-4): 1 least and 4 greatest, total summed score will be used.
Change of antioxidant level | 0 and 40 minutes post snack consumption
  Blood will be collected by finger pricks and change of antioxidant level will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- School of Exercise and Nutritional Sciences, SDSU, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stamper C, Safadi S, Gehr A, Asuncion P, Hong MY. Effects of fresh vs dried mango consumption on satiety and postprandial glucose in healthy adults. Metabol Open. 2023 Jul 18;19:100253. doi: 10.1016/j.metop.2023.100253. eCollection 2023 Sep. PMID 37520177